CLINICAL TRIAL: NCT03701672
Title: A Single-site, Observational Cohort Study to Investigate Predictive Markers of the Effects of Opioid Therapy in Patients With Chronic Pain
Brief Title: Identification of Predictive Markers of the Effects of Opioid Therapy in Patients With Chronic Pain.
Acronym: ABILITY-2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asbjørn Mohr Drewes (Other)
Collaborators: Aleris-Hamlet Hospital (Unknown); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Asbjørn Mohr Drewes, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: ABILITY-2
Record Dates: First submitted 2018-06-19; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Opioid Analgesic Treatment: Chronic paint patients receiving opioid treatment at a Multidisciplinary Pain Center following local SOPs
  Interventions: Other: Opioid Analgesic Treatment

INTERVENTIONS:
Other: Opioid Analgesic Treatment — Opioid treatment is determined, prescribed, modified and discontinued at the sole discretion of the treating physician at each research site; regardless of generic name, manufacturer, constituent components, route of administration, and dosing schedule (including titration and run-in periods).

SUMMARY:
Chronic pain is a significant problem for a large part of the adult population. Opioids are the mainstay of therapy for moderate to severe pain because of their safety, multiple routes of administration, reliability, and effectiveness for all types of pain. However, there is a wide variation in treatment response and a high frequency of side effects associated with the use of opioids. Thus it is important to identify patients who will experience successful pain control with treatment. Unfortunately, as of today no robust objective measures exist for the assessment of the pain-relieving effect of opioids. The pain treatment offered to any given patient is thus largely dependent on the treating physician's experience and the primary pain diagnosis, rather than the characteristics of the individual patient. Unfortunately, this strategy often leads to inadequate treatment, side effects and distress. An implementable clinical tool that can predict and distinguish successful pain control with opioid treatment is therefore warranted.

Quantitative sensory testing (QST) is a method to evaluate the individual pain system. It has been successfully used to describe the problems of individual variation in pain and to predict and measure the responses to an intervention. The investigators recently examined how advanced analyses of QST and pain-related catastrophic thinking could predict opioid response in chronic pain patients whom had not previously received opioid treatment. This study showed that the effect of opioid treatment was predicted by certain pain system responses, catastrophic thinking related to pain and brainwave patterns. The investigators now want to expand on this study by including all patients assigned to opioid treatment by their treating physician. The investigators are also increasing their data collection and using a more elaborate pain system characterization, investigating pain-relevant psychological factors and sleep patter by questionnaires, socio-demographic parameters and collecting descriptive genetic information.

The overall goal of the ABILITY-2 study is to help improve pain diagnostics and treatment by developing an implementable algorithm based on individual patient characteristics to be used in the clinic. The investigators hypothesize that successful pain control with opioids can be predicted before treatment initiation with advanced analyses of QST, pain-related psychological factors and socio-demographic data.

ELIGIBILITY:
Inclusion Criteria:

1. Pain duration ≥ 3 months.
2. Minimum baseline pain intensity ≥ 4 on a 0-10 numerical rating scale (over the past week).
3. Maximum baseline pain intensity < 9 on a 0-10 numerical rating scale (over the past week).
4. Prescribed opioid treatment (ATC: N02)
5. Anticipated to stay on prescribed opioid treatment throughout the study, i.e. >30 days.
6. Anticipated to stay on any concomitant non-opioid treatment throughout the study, i.e. >30 days.
7. Subject may be male or female, age >18 years old.
8. Is willing and able to comply with study procedures as judged by the site investigator.
9. Subject has voluntarily signed and dated the study-specific informed consent form, approved by an Independent Ethics Committee, after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent form must be signed before any study-specific procedures are performed.

Exclusion Criteria:

1. Has a mental incapacity or language barriers precluding adequate understanding of study procedures.
2. Is considered by the site investigator unsuitable to participate in the study for any other reason, for instance due to a significant serious underlying condition.
3. Current alcohol or substance abuse, according to the site investigator's medical judgement.
4. Are suffering from decreased liver function, kidney function, uncontrolled hypertension or currently in treatment with monoamine oxidate (MAO)-inhibitors
5. Is anticipated to undergo a painful procedure(s) (e.g. surgery) during the study, which can interfere with the experience of the chronic pain condition for which the subject is to receive opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants referred tol treatment at a Multidisciplinary Pain Clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in chronic pain assessed by 0-10 numerical rating scale (NRS) scores on the Brief Pain Inventory (BPI) | 30 days
  The absolute and percentage change from baseline in ratings of average pain in the past 24h at Day 30. Of note, a percentage change of ≥30% is considered clinically significant. On the NRS, 0 reflects no pain and 10 reflecs worst pain imaginable in this experimental setup.
Change in health-related quality of life assessed by QLQ-C30 scores | 30 days
  The absolute and percentage change from baseline in ratings of health-related quality of life in the past week at Day 30. A subjectively significant change in QLQ-C30 scores is one that is ≥10 from baseline.The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

SECONDARY OUTCOMES:
Patient Global Impression of Change | 30 days
  Patients impression of change reported as a 7 item assesment of change (1 = much worse and 7 = much better) and the importance of this change (1 = not at all important to 5= extremely important)
The Brief Pain Inventory (BPI) worst pain in the past 24h assessed by 0-10 numerical rating scale (NRS) scores | 30 days
  Change from baseline. On the NRS, 0 reflects no pain and 10 reflecs worst pain imaginable in this experimental setup.
The Brief Pain Inventory (BPI) least pain in the past 24h assessed by 0-10 numerical rating scale (NRS) scores | 30 days
  Change from baseline, On the NRS, 0 reflects no pain and 10 reflecs worst pain imaginable in this experimental setup.
The Brief Pain Inventory (BPI) current pain in the past 24h assessed by 0-10 numerical rating scale (NRS) scores | 30 days
  Change from baseline, On the NRS, 0 reflects no pain and 10 reflecs worst pain imaginable in this experimental setup.
The Brief Pain Inventory (BPI) pain severity in the past 24h assessed by 0-10 numerical rating scale (NRS) scores | 30 days
  Change from baseline, On the NRS, 0 reflects no pain and 10 reflecs worst pain imaginable in this experimental setup.
Severity of Adverse Events | 30 days
  Total score of Adverse Events rated from 1-4 in severity, with 1 being "not at all" and 4 being "Very much". Following adverse events: Constipation, Dry mouth, Nausea/vomiting, Sedation Sweats Bad dreams, Dysphoria/delirium Sleep disturbances, Fatigue, Absent minded, Concentration difficulties, Depressed, Weight gain, Muscle tension, Urination difficulties Ich/Rash, Other

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M Drewes, MD, Study Director — Aalborg University Hospital; Torsten Jonsson, MD, Principal Investigator — Aleris-Hamlet Hospital
Locations (1):
- Aleris-Hamlet Hospital, Ringsted, Denmark

IPD SHARING:
Plan to Share IPD: Undecided